CLINICAL TRIAL: NCT02169661
Title: Lipid Oxidation of Ready Meals: Reformulation With Antioxidant Phytochemicals
Brief Title: Burger and Beetroot Study - Lipid Oxidation Study
Acronym: BABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: HNU 2000
Record Dates: First submitted 2011-07-26; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Oxidative Stress
Keywords: Oxidative stress; Lipid peroxides; Phytochemicals; Ready meals; Beetroot; Blood pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Burger and Beetroot Study (Experimental)
  Interventions: Other: Burger and Beetroot Study

INTERVENTIONS:
Other: Burger and Beetroot Study — 50% fat, 10% beetroot extract

SUMMARY:
Consumption of "ready meals" and other convenience foods are rapidly increasing. However, their nutritional value is problematical. For example, many are high in fats which are potentially oxidisable resulting in the formation of toxic end products. Consequently the aim of this study is to assess whether consumption of "ready meals" rich in certain fats leads to a post-prandial increase in lipid oxidation products in plasma and whether this can be ameliorated by reformulating the meals with natural extracts rich in phytochemicals with potential antioxidant activity in the stomach

DETAILED DESCRIPTION:
Many of these lipid oxidation products such as malondialdehyde are known to be genotoxic and potentially detrimental to health. Consequently the aim of this study is to assess whether consumption of "ready meals" rich in certain fats leads to a post-prandial increase in lipid oxidation products in plasma and whether this can be ameliorated by reformulating the meals with natural extracts rich in phytochemicals with potential antioxidant activity in the stomach.

Diet design requirements:

The basic "ready meal" is a turkey burger consisting of

* 50% fat
* 20% protein
* 30% carbohydrate.

However, there are four experimental forms of the burger.

1. The fat is unsaturated (stripped corn oil)
2. The fat is saturated (lard)
3. The fat is unsaturated and the diet also contains a beetroot extract at a concentration of 10g/100g.
4. The fat is saturated and the diet also contains a beetroot extract at a concentration of 10g/100g.

Beetroot (http://www.kanegrade.com/powders.htm) has been selected for the burger reformulation as it is a Scottish product rich in phytochemicals with potential antioxidant efficacy. An additional benefit may a blood pressure lowering effect. Initial taste tests indicate acceptable palatability.

All other components of the burger are formulated to be as similar as possible.

Fatty acid profiles and the "basic eight" used on food labels will be determined on the diets. Susceptibility of the diets to oxidise will be assessed using RANCIMAT.

Ready Meal Intervention:

This will be a latin square format whereby each volunteer consumes 4 treatments on separate occasions. This is a powerful design to assess whether incorporation of phytochemicals from Scottish products improves the health benefits of processed food as each volunteer acts as his/her own control. Volunteers will be randomly allocated to four groups

* Treatment A High polyunsaturated (PUFA) ready meal (ie. burger)
* Treatment B High saturated (SFA) fat ready meal
* Treatment C High PUFA ready meal incorporating food extract
* Treatment D High SFA ready meal incorporating food extract

There will be a washout period of at least 7 days between each treatment.

Volunteers:

Healthy volunteers aged 21 to 60 years will be recruited and attend HNU having fasted from 22.00h the previous evening on four test days. On arrival, they will be asked to provide a urine sample. The volunteers will then have a cannula inserted by a trained nurse and an initial baseline blood sample will be taken (volume 10 ml). The subjects will then be asked to consume the assigned breakfast within a 15 minute period. Water will be provided. Volunteers will then be requested to provide 10ml blood samples at 1h, 2h, 4h and 6h and 24 hrs. A 24 hr urine sample also will be obtained, starting the day of the test day. Blood pressure will be recorded at each time point.

Volunteers will not be included if they

* Are taking any medicines prescribed by their GP
* Have a known allergy to beetroot
* Are vegetarian or vegan
* Regularly take nutritional supplements
* Have given a large blood donation in last three months

ELIGIBILITY:
Inclusion Criteria:

* No diagnosed clinical condition

Exclusion Criteria:

Are taking any medicines prescribed by their GP Have a known allergy to beetroot Are vegan Regularly take nutritional supplements Have given a large blood donation in last three months

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Lipid peroxides | up to 24 hours
  Indices of oxidised lipids in plasma

SECONDARY OUTCOMES:
Blood pressure | up to 24 hours
  Systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Garry G Duthie, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Human Nutrition Unit, Rowett Institute of Nutrition and Health, Aberdeen, Scotland, United Kingdom